CLINICAL TRIAL: NCT03664908
Title: Detection of Anti-glomerular Basement Membrane Antibodies (Anti-GBM): a Promising Biomarker for Lupus Nephritis (LN) Screening in Systemic Lupus Erythematosus (SLE) Patients?
Brief Title: Detection of Anti-glomerular Basement Membrane Antibodies (Anti-GBM): a Promising Biomarker for Lupus Nephritis (LN)?
Acronym: GOODLUPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PO18049
Record Dates: First submitted 2018-07-23; First posted 2018-09-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2020-06

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; systemic lupus erythematosus; anti-glomerular basement membrane disease anti-GBM antiboby
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — Fluorescent Antibody Technique, Indirect; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- serum samples of SLE patients without LN (Experimental): 100 serum samples coming from systemic lupus erythematosus (SLE) patients without lupus nephritis (LN).
  Interventions: Other: Detection of circulating anti-GBM antibodies (using chemiluminescence method and indirect immunofluorescence (IIF) method).
- serum samples of Lupus nephritis (LN) patients (Experimental): 100 serum samples coming from systemic lupus erythematosus(SLE) patients with lupus nephritis (LN)
  Interventions: Other: Detection of circulating anti-GBM antibodies (using chemiluminescence method and indirect immunofluorescence (IIF) method).
- healthy voluntary blood donors (control group) (Experimental): 100 serum sample coming from 100 healthy voluntary blood donors (provided by Regional blood center of Reims). This arm will be our control group.
  Interventions: Other: Detection of circulating anti-GBM antibodies (using chemiluminescence method and indirect immunofluorescence (IIF) method).

INTERVENTIONS:
Other: Detection of circulating anti-GBM antibodies (using chemiluminescence method and indirect immunofluorescence (IIF) method). — biological detection of circulating anti-GBM antibodies (using chemiluminescence method and indirect immunofluorescence (IIF) method) in three serum samples groups, coming from SLE patients (having Lupus Nephritis or not) and in a control group.

SUMMARY:
Introduction and background :

Glomerulonephritis and auto-immune diseases are often associated. Lupus nephritis (LN) is one of the major clinical manifestations of systemic lupus erythematosus (SLE) which have a severe impact on prognosis. This complication is a real challenge for clinicians because of insidious-onset and no predictable relapses. Biomarker use is therefore essential, but conventional biomarkers such as proteinuria have poor sensivity and low specificity to predict LN occurrence, and new more reliable biomarkers (genetic, epigenetic or protein biomarkers) are difficult to use for daily medical practice.

Anti-glomerular membrane basement disease (anti-GBM disease) is a rare (0.5 to 1/millions of inhabitants) and severe illness, characterised by rapidly progressive glomerulonephritis, pulmonary haemorrhage and the presence of anti-GBM antibodies, which are highly sensible (100%) and specific (92-100%) of this condition

. Our experience and literature review

In our department of internal medicine, we report one case of anti-GBM glomerulonephritis associated to an active SLE. After literature review, we note the following studies:

* some similar association cases had been reported.
* In 2006, a Chinese cohort study highlighted important rates of anti-GBM antibodies, in serum samples from patients with SLE (14 positives/157patients (8.9%) using ELISA method). Moreover, every SLE patient with positive circulating anti-GMB antibodies LN and a severer SLE (with significantly more anemias, pulmonary hemorrhage). According to histological data's, they also had more important kidney damages (10/14 had necrotizing crescentic glomerulonephritis lesions and 5/14 fulfil criteria's for anti-GBM disease diagnosis).
* We also note that some authors published experimental studies showing that immunological and genetic links exist between LN and anti-GBM disease, which could explain this association.

  3. Main Hypothesis: Based on these findings, we suspect that detection of significant levels of circulating anti-GBM antibodies may be more frequent in SLE followed patients than in general population, and that it could be an interesting biomarker of LN in patient with SLE.

  4. Objectives First objective: based on 2 SLE patient groups (one having lupus nephritis and the other without it) we would like to compare the ratio of positive anti-GBM antibodies in each group, expecting a higher rate in SLE patients with LN.

Second objective: will be to study the positive anti-GBM group patients in their clinical aspects, serological features and renal characteristics, in this SLE population.

5. Materials and methods We suggest a retrospective analytic transversal controlled study, based on serum samples from the Lupus Biobank of Upper Rhine (LBBR project), and based on serum samples from healthy voluntary blood donors (control group). We will then perform tests in each serum sample group in our immunology laboratory and compare the ratio of positive anti-GBM in each arm.

DETAILED DESCRIPTION:
Introduction and context :

Glomerulonephritis and auto-immune diseases are often associated. Lupus nephritis (LN) is one of the major clinical manifestations of systemic lupus erythematosus (SLE) which have a severe impact on prognosis. This complication is a real challenge for clinicians because of insidious-onset and no predictable relapses. Biomarker use is therefore essential, but conventional biomarkers such as proteinuria, glomerular filtration rate, urine sediments, anti-dsDNA antibodies and complement levels, have poor sensivity and low specificity to predict LN occurrence, and new more reliable biomarkers (such as genetic, epigenetic or protein biomarkers) are difficult to use for daily medical practice , .

Anti-glomerular membrane basement disease (anti-GBM disease) is a rare (0.5 to 1/millions of inhabitants , ) and severe illness , , characterised by rapidly progressive glomerulonephritis, pulmonary haemorrhage and the presence of anti-GBM antibodies, which are highly sensible (100%) and specific (92-100%) of this condition .

In our department of internal medicine, one case of Goodpasture glomerulonephritis associated to an active SLE has been reported , and after searching data in literature, we note the following studies:

* some similar cases were reported such as a case of pulmonary hemorrhage and positive anti-GBM in SLE , or a case of anti-GBM disease and LN presenting as pulmonary-renal syndrome .
* In 2006, a Chinese cohort study highlighted an elevated prevalence of anti-GBM antibodies, in serum samples from patients with SLE (14 positives/157patients (8.9%) with ELISA method). Moreover, every patient with positive anti-GMB antibodies had LN and a severer SLE (with more anemias, pulmonary hemorrhage). They also suffered from more important kidney disease. In fact, in histological criteria's, 10/14 had necrotizing crescentic glomerulonephritis lesions and 5/14 had a real diagnosis of Goodpasture disease.
* We also note that some authors have already studied pathogenesis of this association (whether immunological explanations , genetics links , ).

  3. Main Hypothesis: Based on these findings, we suspect that detection of positive circulating anti-GBM antibodies may be more frequently positive in SLE followed patients (than in general population) and that it could be an interesting screening biomarker for LN.

  4. Objectives First objective: based on 2 SLE patient groups (one having lupus nephritis and another without it) we would like to compare the ratio of positive anti-GBM antibodies in each group, expecting a higher rate in SLE patients with LN.

Second objective: to study positive anti-GBM patients in their clinical aspects, serological features and renal characteristics, in this SLE population.

5. Materials and methods We suggest a retrospective analytic transversal controlled study, based on serum samples from the Lupus Biobank of Upper Rhine (LBBR project), and on serum samples from healthy voluntary blood donors (control group).

Regarding the use of LBBR Lupus Biobank, our project has already been accepted by scientific committee.

After group randomization, Cryo-conserved SLE serum samples will be transferred by specialized transporter service, from Strasbourg biobank, to the immunology laboratory department in Reims University Hospital center, to perform anti-GBM tests.

Concerning healthy serum sample recruitment, Regional blood center of Reims will systematically suggest to voluntary blood donors to participate. If they agree, they will receive an extended information about the study, and after written consent, a tube sample will be collected.

6. Population The statistic calculation led to the need of 200 SLE sera (100 patients in each group). Thus, we will use : 100 serum samples coming from lupus biobank LBBR patients without lupus nephritis, and 100 serum samples of patients with systemic lupus erythematosus and lupus nephritis.

We will also use 100 serum samples of voluntary blood donors.

7. Experimental project Anti-GBM antibodies detection in serums will be performed by an automatized chemiluminescent method, using a commercial test kit. In case of positivity, same serum will be tested second time to confirm the result, and then controlled by another method using indirect immunofluorescence (IIF) in frozen sections of primate kidney, covering the reaction areas of a BIOCHIP slide (reference method).

According to our immunology laboratory department, we need 600μl of serum per patient to be able to perform all the tests. According to the manufacturer's instruction, the optimum cut-off value for positivity in chemiluminescence method will be set at 20CU/mL.

8. Data analysis Primary endpoint: proportion of positive anti-MBG antibodies, will be estimated in each group (with and without lupus nephritis) by a Chi-2 test or an exact test of Fisher (depending on test validity conditions).

Secondary endpoint: clinical, serological and renal features of anti-GBM positives patients, will be compared to negatives, using tests adapted to the distribution of each variable.

9. Expected results and future prospects

* We expect a higher frequency of positive circulating anti-GBM antibodies in patients with LN compared to the SLE control group and to healthy control group.
* Whether this research was positive, another larger study could show the interest of anti-GBM antibodies as a predictive biomarker of LN, and as a prognostic biomarker of SLE.

ELIGIBILITY:
Inclusion Criteria:

* serum samples coming from LBBR lupus biobank (diagnosis of lupus according ACR criteria or diagnosis of lupus nephritis according to ISN/RPS2003) or serum sample coming from healthy bload donor volunters
* having signed the informed consent

Exclusion Criteria:

* diagnosis of lupus nephritis and having a beginning kidney disease (every class I and II of WHO classification and class I or II of ISN/RPS classification)
* lack of data regarding kidney histology on clinical LBBR file
* minor healthy blood donor
* healthy blood donor volunters with auto immune disease, or kidney disease, or chronic renal failure or taking immunosuppressive or immunomodulatory therapy or with history of cutaneous lupus or SLE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Percentage of serum with anti GBM positivity | Day 0
  circulating antibody rates higher than 20 cu/mi using chemiluminescence

SECONDARY OUTCOMES:
Description of clinical features of patients | Day 0
  as gender, ethnical group and mean age of patients
Description of SLE characteristics | Day 0
  as age of disease onset, ACR criteria in patients with and without anti GBM positivity
Description of immunological characteristics of patients with anti GBM positivity | Day 0
  presence of other auto immune disease, lupus anticoagulant, false positive syphilis test anticandidipid
Description of renal characteristics of patient with anti GBM positivity | Day 0
  presence kidney disease or significant proteinurie or hemaluria or pyuria or urinary casts and kidney histology

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Bourse Chalvon N, Orquevaux P, Giusti D, Gatouillat G, Tabary T, Tonye Libyh M, Chrusciel J, Drame M, Stockton-Bliard G, Amoura Z, Arnaud L, Lorenz HM, Blaison G, Bonnotte B, Magy-Bertrand N, Revuz S, Voll RE, Hinschberger O, Schwarting A, Pham BN, Martin T, Pennaforte JL, Servettaz A. Absence of Anti-Glomerular Basement Membrane Antibodies in 200 Patients With Systemic Lupus Erythematosus With or Without Lupus Nephritis: Results of the GOODLUPUS Study. Front Immunol. 2020 Dec 14;11:597863. doi: 10.3389/fimmu.2020.597863. eCollection 2020. PMID 33381119